CLINICAL TRIAL: NCT01723007
Title: Modifications of Body Weight and Plasma Lipids With Diet Added of Fruits: Randomized Clinical Trial in Overweight Women
Brief Title: Weight Loss Associated With the Consumption of Apple
Acronym: NCTAPPLEBR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Amazonas (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Associação Brasileira de Produtores de Maçã - ABPM (Unknown); Hospital Universitario Pedro Ernesto (Other); Universidade do Estado do Rio de Janeiro - UERJ (Unknown)
Responsible Party: Principal Investigator, Maria Conceição de Oliveira, Doctor; Associate Professor of Epidemiology, Universidade Federal do Amazonas
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: ABPM_NCT_APPLE_BR1999
Record Dates: First submitted 2012-10-09; First posted 2012-11-07 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Hypercholesterolemia; Overweight
Keywords: Weight loss; cholesterol
MeSH Terms: conditions — Hypercholesterolemia; Overweight; Weight Loss | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Other: Apple (Experimental): Women were supplemented with apples. Sixteen women were asked to ingest three apple daily between meals ( approximately 120g kcal) between meals (breakfast, lunch and dinner).
  Interventions: Other: Supplement
- Other: oatmeal cookies (Active Comparator): A another group with nineteen women were asked to ingest three oatmeal cookies a day, approximately 60g and similar caloric content to experimental group (approximately 120 kcal) between meals (breakfast, lunch and dinner).
  Interventions: Other: Supplement
- Other: Pear (Active Comparator): Women were supplemented with pear. Sixteen women were asked to ingest daily three pears (approximately 120 kcal) between meals daily (breakfast, lunch and dinner).
  Interventions: Other: Supplement

INTERVENTIONS:
Other: Supplement — The arms were assigned to receive the supplements and followed for 10 weeks. Every two weeks, the women returned to the clinic for evaluation biochemical, haemogram, anthropometric, bioimpedance, blood pressure and dietary. Weekly, returned to receive the supplements in a sealed box. They received guidance not to disclose what food were receiving the service if he found other women who also participated in the study.
  Other Names: Dietary supplement

SUMMARY:
The study was designed to answer the primary question: the consumption of one apple three times daily between meals reduces serum levels of cholesterol above 240 mg/dL in overweight women? The second and important hypothesis was designed for evaluate the reduction in body weight by intakes of fruits. Therefore, the increased consumption of apples could displace the consumption of other foods and promoting satiety and input significant reduction in body weight compared to other fruit (Pear) of similar nutritional composition or food (cookies) made from oats with fiber and total calories similar to those observed in these fruits. To demonstrate the effectiveness of these supplements we used a clinical trial with three arms (apple, pear and oatmeal cookies).

DETAILED DESCRIPTION:
The basic proposal of this research was to study the effect of apple consumption as dietary treatment of plasma lipids and weight loss. To assess the effect of apple adding in diet, first was necessary to standardize the total number of meals, since the serum cholesterol level is influenced by this variation. Thus, in the run-in period of the study the researchers stabilized the number of meals. The participants increased the number of meals with introduction of three supplements daily.

A possible physiological basis for the hypothesis of a protective effect of apples on serum cholesterol and body weight would be their fiber composition, so the study presents a comparison arm for the consumption of dietary fiber adjusted for total calories (oatmeal cookies). However, another possible physiological factor could be the energy density of foods. Energy density is an important determinant of energy consumption because a high intake of a diet low energy-dense food, such as fruits, makes excessive energy consumption more difficult, and few studies have been conducted on satiety and weight control and serum cholesterol. Recently (2012) discovered the presence on the apple peel a substance named ursolic acid that showed the effect in reducing body weight.

Previous studies have observed a reduction in cholesterol levels associated with consumption of apple and for to test this hypothesis, as well as weight reduction, a randomized clinical trial study with three arms where the apple was compared with an equal amount of fiber and total calories by eating oatmeal cookies and other fruit (pear).

We postulated that, if a group receive an other fruit could be excluding the possibility of the effect being attributed to the increased consumption of fruits displacing other foods and not apple effect. The pear was chosen due to its percentage of the nutritional components similar the apple. Before beginning the survey raised the consumption of apple in Brazil to assess the feasibility of such a study, if we confirmed the hypothesis of a protective effect. The apple consumption in Brazil increased in recent years. This trend was driven by the increased supply of fruit and reduction of food prices in general. Still in the pilot study survey we tested the acceptance of the introduction of three fruits in the diet of participants. The majority of the population accepted without problems to ingest three fruits daily. Our initial hypothesis was that fruit consumption in low-income populations would be low, which was confirmed. To ensure increased consumption of fruits, these were purchased and delivered to the participants, along with transportation vouchers, weekly. The oat cookies were also produced by the staff and offered at no cost to the participants. The frequency of the number of daily meals was low in the study population at baseline: 3.8 meals per day and could encourage major changes in lipid metabolism, associated to the frequency of meals. Then, the number of meals was increased to six meals a day, including breakfast, lunch, dinner and three snacks between meals and supplement: apple, pear or oat cookies. The dietary prescription was based on the eating habits of participants at baseline, changing only the number of meals and by introduce fruits or biscuits during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women with hypercholesterolemia,
* Body Mass Index: IMC > 25 Kg/m2,
* No smoking,
* Between 30 to 50 years;
* Report like apple and pear.

Exclusion Criteria:

* Changes in diet in the last 6 months,
* Making use of controlled medication,
* Pregnant or lactating women.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 1999-08; Primary Completion 2000-06 (Actual); Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Cholesterol | Ten weeks
  The plasma cholesterol was evaluated every two weeks . After 10 weeks of follow-up the consumption of three apple reduced serum cholesterol, but was not statistically significant.
Body weight | Ten weeks
  The body weight was evaluated every two weeks.

SECONDARY OUTCOMES:
Increased triglycerides | Ten weeks
  Adherence to fruit consumption by participants was evaluated through the changes of serum triglycerides During 4 weeks of follow up.

OTHER OUTCOMES:
Caloric and nutrient intakes | Ten weeks
  To assess adherence to diet and supplements (apple, pear or oat cookies) was used food records twice a week and on weekends.
Nutritional Composition of Diet | Ten weekes
  Food frequency questionnaire was used for analyzing of fiber, calorie content and caloric density on body weight during 10 weeks of follow up. The results were published.
Frequency of meals | Ten weeks
  The frequency of meals daily changes in 10 weeks of follow up were analyzed
Blood Biochemistry | Ten weeks
  The possibility of changes in blood biochemistry for serum urea and serum creatinine, glucose,insulin, haemogram, and lipids fractions during 10 weeks of follow up were analysed. These fractions were not analyzed.
Anthropometry | Ten weeks
  Circumferences (arm, wrist, waist and abdominal), skinfold thickness (biceps, triceps, subscapular, abdominal and calf). Sitting height and standing height in 10 weeks of follow up. Measures are yet to be analyzed.
Blood pressure | Ten weeks
  Blood pressure was evaluated every two weeks during 10 weeks of follow up. The outcomes were not disclosed.
Bioelectrical Impedance | Ten weeks
  The bioelectrical impedance (inductance, resistance) was evaluated to access the phase angle during 10 weeks of follow up. Measures are yet to be analyzed.
Urinalysis | Ten weeks
  Urine analysis was performed to monitor renal function in the three groups (apple, pear and oatmeal cookies), verify changes in urine color and concentration during 10 weeks of follow up. The measures are still being considered.

CONTACTS AND LOCATIONS:
Overall Officials: Maria C De Oliveira, Doctor, Principal Investigator — Universidade Federal do Amazonas
Locations (2):
- Brazil (2):
  - Department of Public Health-DSC, School of Medicine-FM, University of Aamazon-UFAM, Manaus, Amazonas
  - Department of Public Health-DSC-FM School of Medicine, Federal University of Amazon-UFAM, Manaus-AM, Amazonas

REFERENCES:
- [Background] Raynor HA, Looney SM, Steeves EA, Spence M, Gorin AA. The effects of an energy density prescription on diet quality and weight loss: a pilot randomized controlled trial. J Acad Nutr Diet. 2012 Sep;112(9):1397-1402. doi: 10.1016/j.jand.2012.02.020. Epub 2012 May 9. PMID 22575072
- [Background] Vergnaud AC, Norat T, Romaguera D, Mouw T, May AM, Romieu I, Freisling H, Slimani N, Boutron-Ruault MC, Clavel-Chapelon F, Morois S, Kaaks R, Teucher B, Boeing H, Buijsse B, Tjonneland A, Halkjaer J, Overvad K, Jakobsen MU, Rodriguez L, Agudo A, Sanchez MJ, Amiano P, Huerta JM, Gurrea AB, Wareham N, Khaw KT, Crowe F, Orfanos P, Naska A, Trichopoulou A, Masala G, Pala V, Tumino R, Sacerdote C, Mattiello A, Bueno-de-Mesquita HB, van Duijnhoven FJ, Drake I, Wirfalt E, Johansson I, Hallmans G, Engeset D, Braaten T, Parr CL, Odysseos A, Riboli E, Peeters PH. Fruit and vegetable consumption and prospective weight change in participants of the European Prospective Investigation into Cancer and Nutrition-Physical Activity, Nutrition, Alcohol, Cessation of Smoking, Eating Out of Home, and Obesity study. Am J Clin Nutr. 2012 Jan;95(1):184-93. doi: 10.3945/ajcn.111.019968. Epub 2011 Dec 14. PMID 22170373
- [Background] Ello-Martin JA, Roe LS, Ledikwe JH, Beach AM, Rolls BJ. Dietary energy density in the treatment of obesity: a year-long trial comparing 2 weight-loss diets. Am J Clin Nutr. 2007 Jun;85(6):1465-77. doi: 10.1093/ajcn/85.6.1465. PMID 17556681
- [Background] Ello-Martin JA, Ledikwe JH, Rolls BJ. The influence of food portion size and energy density on energy intake: implications for weight management. Am J Clin Nutr. 2005 Jul;82(1 Suppl):236S-241S. doi: 10.1093/ajcn/82.1.236S. PMID 16002828
- [Background] Rolls BJ, Roe LS, Beach AM, Kris-Etherton PM. Provision of foods differing in energy density affects long-term weight loss. Obes Res. 2005 Jun;13(6):1052-60. doi: 10.1038/oby.2005.123. PMID 15976148
- [Background] Singh RB, Niaz MA, Bishnoi I, Singh U, Begum R, Rastogi SS. Effect of low energy diet and weight loss on major risk factors, central obesity and associated disturbances in patients with essential hypertension. J Hum Hypertens. 1995 May;9(5):355-62. PMID 7623373
- [Background] Lin J, Fung TT, Hu FB, Curhan GC. Association of dietary patterns with albuminuria and kidney function decline in older white women: a subgroup analysis from the Nurses' Health Study. Am J Kidney Dis. 2011 Feb;57(2):245-54. doi: 10.1053/j.ajkd.2010.09.027. PMID 21251540
- [Background] Sacks FM, Appel LJ, Moore TJ, Obarzanek E, Vollmer WM, Svetkey LP, Bray GA, Vogt TM, Cutler JA, Windhauser MM, Lin PH, Karanja N. A dietary approach to prevent hypertension: a review of the Dietary Approaches to Stop Hypertension (DASH) Study. Clin Cardiol. 1999 Jul;22(7 Suppl):III6-10. doi: 10.1002/clc.4960221503. PMID 10410299
- [Background] Lin PH, Windhauser MM, Plaisted CS, Hoben KP, McCullough ML, Obarzanek E. The Linear Index Model for establishing nutrient goals in the Dietary Approaches to Stop Hypertension trial. DASH Collaborative Research Group. J Am Diet Assoc. 1999 Aug;99(8 Suppl):S40-4. doi: 10.1016/s0002-8223(99)00415-0. PMID 10450293
- [Background] Appel LJ, Moore TJ, Obarzanek E, Vollmer WM, Svetkey LP, Sacks FM, Bray GA, Vogt TM, Cutler JA, Windhauser MM, Lin PH, Karanja N. A clinical trial of the effects of dietary patterns on blood pressure. DASH Collaborative Research Group. N Engl J Med. 1997 Apr 17;336(16):1117-24. doi: 10.1056/NEJM199704173361601. PMID 9099655
- [Background] Hyson D, Studebaker-Hallman D, Davis PA, Gershwin ME. Apple juice consumption reduces plasma low-density lipoprotein oxidation in healthy men and women. J Med Food. 2000 Winter;3(4):159-66. doi: 10.1089/jmf.2000.3.159. PMID 19236172
- [Background] Sable-Amplis R, Sicart R. Hepatic acylcoenzyme A:cholesterol acyltransferase activity is low in hamsters fed apples in addition to a standard diet. Ann Nutr Metab. 1993;37(1):1-7. doi: 10.1159/000177742. PMID 8470868
- [Background] Sable-Amplis R, Sicart R, Dupouy D. Hepatic cholesterogenesis and cholesterol 7 alpha-hydroxylase activity in hamsters fed diets enriched with pectins and/or cholesterol. Ann Nutr Metab. 1987;31(1):61-8. doi: 10.1159/000177249. PMID 3827206
- [Background] Chai SC, Hooshmand S, Saadat RL, Payton ME, Brummel-Smith K, Arjmandi BH. Daily apple versus dried plum: impact on cardiovascular disease risk factors in postmenopausal women. J Acad Nutr Diet. 2012 Aug;112(8):1158-68. doi: 10.1016/j.jand.2012.05.005. PMID 22818725
- [Result] de Oliveira MC, Sichieri R, Venturim Mozzer R. A low-energy-dense diet adding fruit reduces weight and energy intake in women. Appetite. 2008 Sep;51(2):291-5. doi: 10.1016/j.appet.2008.03.001. Epub 2008 Mar 7. PMID 18439712
- [Result] Conceicao de Oliveira M, Sichieri R, Sanchez Moura A. Weight loss associated with a daily intake of three apples or three pears among overweight women. Nutrition. 2003 Mar;19(3):253-6. doi: 10.1016/s0899-9007(02)00850-x. PMID 12620529